CLINICAL TRIAL: NCT04167904
Title: Biomarkers in Patients Hospitalized With Suspected Acute Myocardial Infarction
Acronym: BIOMAC
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/648
Record Dates: First submitted 2018-09-03; First posted 2019-11-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Infarction, Acute
Keywords: Troponin I; Myocardial Infarction; Sensitivity and Specificity; Receiver operation characteristics curve; Biomarkers
MeSH Terms: conditions — Myocardial Infarction; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, lithium heparin plasma and EDTA blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The concentration of troponins in plasma is used for diagnosing acute myocardial infarction. Different types of heart-specific troponins can be measured and with different analytical methods. The primary aim of this study is to evaluate the diagnostic characteristics of a new analytical method for measuring troponin I in diagnosing acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized at St. Olavs hospital
* blood sampled for troponin analysis due to suspicion of acute myocardial infarction without ST-elevations on ECG less than 4 hours after admitted to the hospital

Exclusion Criteria:

* residency outside Norway
* does not understand Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to St. Olavs Hospital (Trondheim University Hospital) with suspected acute myocardial infarction without ST-elevations on ECG (NSTEMI).
Sampling Method: Non-Probability Sample
Enrollment: 4446 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Acute myocardial infarction according to the 4th universal definition of myocardial infarction | Before discharge from hospital, a median of 2 days
  Metric: Yes/No

SECONDARY OUTCOMES:
Days between hospital discharge and death | Within 30 days after hospital discharge
  Metric: Days. The secondary outcome measures will be combined into a composite endpoint reflecting the time between hospital admission and the first secondary outcome measure
Days between hospital discharge and acute myocardial infarction according to the 4th universal definition of myocardial infarction | Within 30 days after hospital discharge
  Metric: Days.
Days between hospital discharge and coronary revascularization | Within 30 days after hospital discharge
  Metric: Days

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Mikkelsen, MD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided